CLINICAL TRIAL: NCT00769496
Title: A Long-term, Open Label Extension, Non-controlled Study to Assess the Efficacy and Safety of BAY 77-1931 (Lanthanum Carbonate) for Hyperphosphatemia in Patients Undergoing Hemodialysis
Brief Title: BAY 77-1931 Long-term Extension From Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Yakuhin Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11551
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY 77-1931

INTERVENTIONS:
Drug: BAY 77-1931 — Lanthanum Carbonate (BAY 77-1931)

SUMMARY:
A long-term study of BAY77-1931 (lanthanum carbonate) for hyperphosphatemia in patients undergoing hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Undergoing hemodialysis 3 times per week for chronic renal failure for the previous 3 consecutive months at least

Exclusion Criteria:

* Pre-dialysis serum phosphate levels of 10.0mg/dL during the washout period

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Changes in pre-dialysis serum phosphate levels | Every 4 weeks

SECONDARY OUTCOMES:
Achievement rate of the target predialysis serum phosphate levels (3.5 mg/dL and 5.5 mg/dL) | Every 4 weeks
Changes in corrected serum calcium level | Every 4 weeks
Changes in the product of serum calcium and phosphate | Every 4 weeks
Changes in serum intact-PHT levels | Every 4 weeks
Changes in bone metabolism markers | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- Japan (12):
  - Toyohashi, Aichi-ken
  - Yatomi, Aichi-ken
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Narita, Chiba
  - Sakura, Chiba
  - Hiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Kochi, Kochi
  - Okayama, Okayama-ken
  - Suita, Osaka
  - Tokushima, Tokushima